CLINICAL TRIAL: NCT03998696
Title: Comparison Between Two Regimens of Chemotherapy Concurrent With Radiotherapy in Locally Advanced Head and Neck Cancer
Brief Title: An Experimental Study to Compare Treatment Response and Toxicities of Concurrent Chemoradiation With Weekly Cisplatin and Three Weekly Cisplatin in Locally Advanced Head and Neck Cancer.
Acronym: HNC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Ishtiaq-Ur-Rahim, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2017/1577; 2017/311 (Other: NICRH)
Record Dates: First submitted 2019-06-22; First posted 2019-06-26 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Locally advanced; Head and Neck Cancer; Concurrent; Weekly Cisplatin; Three weekly Cisplatin; Radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weekly Cisplatin (Active Comparator): Inj. Cisplatin 40 mg /m2 intravenous infusion delivered concurrently with radiotherapy on a weekly basis.
  Interventions: Drug: Cisplatin 40 mg/m2
- Three weekly Cisplatin (Experimental): Inj. Cisplatin 100 mg/m2 intravenous infusion delivered on a three weekly basis on days 1, 22 and 43 delivered concurrently with radiotherapy.
  Interventions: Drug: Cisplatin 100 mg/m2

INTERVENTIONS:
Drug: Cisplatin 40 mg/m2 — Cisplatin 40 mg/m2, weekly, concurrent with Radiotherapy
  Arms: Weekly Cisplatin
Drug: Cisplatin 100 mg/m2 — Cisplatin 100 mg/m2, three weekly, concurrent with Radiotherapy
  Arms: Three weekly Cisplatin

SUMMARY:
The aim of this study is to compare treatment responses and toxicities of concurrent chemo-radiation with weekly and three weekly Cisplatin in locally advanced Head & Neck Cancer. Half of the participants received Cisplatin (40 mg/m2) weekly with radiotherapy, while the other half received Cisplatin (100 mg/m2) thrice weekly with radiotherapy. Radiotherapy continued five days per week for six and half weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proved, previously untreated, Squamous cell carcinoma of head & neck
* Stages III to IVB

Exclusion Criteria:

* Patients with history of prior chemotherapy or radiotherapy to the head and neck region.
* Initial surgery (excluding diagnostic biopsy) of the primary site.
* Patients with synchronous primaries.
* Those who are not willing to be included in the study.
* Pregnant or lactating woman.
* Serious medical illness
* Prisoners.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Loco-regional tumor control after completion of treatment | 6 months
  Response Evaluation Criteria in Solid Tumors was used to measure outcome:
  1. Complete response (CR): Disappearance of all target lesions.
  2. Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  3. Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions.
  4. Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Treatment related toxicities during and after treatment | 8 months
  National Cancer Institute's Common Terminology Criteria for Advanced Events (version 4.03) was used measure toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Sarwar Alam, MBBS, Mphil, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Access Criteria: To request an electronic copy send email to dr.iurahim@gmail.com

REFERENCES:
- [Background] Adelstein DJ, Li Y, Adams GL, Wagner H Jr, Kish JA, Ensley JF, Schuller DE, Forastiere AA. An intergroup phase III comparison of standard radiation therapy and two schedules of concurrent chemoradiotherapy in patients with unresectable squamous cell head and neck cancer. J Clin Oncol. 2003 Jan 1;21(1):92-8. doi: 10.1200/JCO.2003.01.008. PMID 12506176
- [Background] Geeta SN, Padmanabhan TK, Samuel J, Pavithran K, Iyer S, Kuriakose MA. Comparison of acute toxicities of two chemotherapy schedules for head and neck cancers. J Cancer Res Ther. 2006 Jul-Sep;2(3):100-4. doi: 10.4103/0973-1482.27584. PMID 17998687
- [Background] Guan J, Zhang Y, Li Q, Zhang Y, Li L, Chen M, Xiao N, Chen L. A meta-analysis of weekly cisplatin versus three weekly cisplatin chemotherapy plus concurrent radiotherapy (CRT) for advanced head and neck cancer (HNC). Oncotarget. 2016 Oct 25;7(43):70185-70193. doi: 10.18632/oncotarget.11824. PMID 27602493
- [Background] Ho KF, Swindell R, Brammer CV. Dose intensity comparison between weekly and 3-weekly Cisplatin delivered concurrently with radical radiotherapy for head and neck cancer: a retrospective comparison from New Cross Hospital, Wolverhampton, UK. Acta Oncol. 2008;47(8):1513-8. doi: 10.1080/02841860701846160. PMID 18607863
- [Background] Jacinto JK, Co J, Mejia MB, Regala EE. The evidence on effectiveness of weekly vs triweekly cisplatin concurrent with radiotherapy in locally advanced head and neck squamous cell carcinoma (HNSCC): a systematic review and meta-analysis. Br J Radiol. 2017 Nov;90(1079):20170442. doi: 10.1259/bjr.20170442. PMID 29053029
- [Background] Lee JY, Sun JM, Oh DR, Lim SH, Goo J, Lee SH, Kim SB, Park KU, Kim HK, Hong DS, Kim JS, Kim SG, Yi SY, Yun HJ, Hyun MS, Kim HJ, Jung SH, Park K, Ahn YC, Ahn MJ. Comparison of weekly versus triweekly cisplatin delivered concurrently with radiation therapy in patients with locally advanced nasopharyngeal cancer: A multicenter randomized phase II trial (KCSG-HN10-02). Radiother Oncol. 2016 Feb;118(2):244-50. doi: 10.1016/j.radonc.2015.11.030. Epub 2015 Dec 17. PMID 26705681
- [Background] Tsan DL, Lin CY, Kang CJ, Huang SF, Fan KH, Liao CT, Chen IH, Lee LY, Wang HM, Chang JT. The comparison between weekly and three-weekly cisplatin delivered concurrently with radiotherapy for patients with postoperative high-risk squamous cell carcinoma of the oral cavity. Radiat Oncol. 2012 Dec 18;7:215. doi: 10.1186/1748-717X-7-215. PMID 23245290
- See also: Global Cancer Observatory (GLOBOCAN), 2018. — http://gco.iarc.fr/today/fact-sheets-populations